# **Title:** Comparison Between the Use of Music and Relaxation Training on Craving Alcohol in Patients with Alcohol Dependence Syndrome:

A Pilot Study

**NCT No:** NCT04351217

By Shradha Chandrasekar

Date: 16 January, 2019



## Department of Psychiatry, Kasturba Medical College, Mangalore, Karnataka, India

NCT No.: NCT04351217

Comparison Between the Use of Music and Relaxation Training on Craving Alcohol in Patients with Alcohol Dependence Syndrome:

A Pilot Study

By Shradha Chandrasekar

Under the Guidance of: Dr Keshava Pai,
Professor and Head, Dept of Psychiatry
KMC Mangalore

## **Table of Contents**

| S. No. | Topic | Page No |
|--------|------------------------|---------|
| 1. | Introduction | 3 |
| 2 | Review of Literature | 9 |
| 3 | Rationale of the Study | 12 |
| 4 | Need for the Study | 13 |
| 5 | Methodology | 14 |
| 6. | Procedure | 17 |
| 7 | References | 20 |
| 8 | Appendix | 24 |

#### Introduction

#### **Alcohol Dependence Syndrome (ADS)**

A cluster of physiological, behavioural, and cognitive phenomena in which the use of a substance (here, alcohol) or a class of substances takes on a much higher priority for a given individual than other behaviours that once had greater value.

Diagnostic guidelines include

- 1. Strong desire or sense of compulsion to take substance;
- 2. Difficulties in controlling substance-taking behaviour in terms of its onset, termination, or levels of use;
- 3. A physiological withdrawal state

(Includes symptoms experienced in the Head: headaches, dizziness; Chest: Chest tightness, difficulty breathing; Heart: Racing heart, skipped beats, palpitations; GI: Nausea, vomiting, diarrhoea, stomach aches; Muscles: Muscle tension, twitches, tremors, shakes, muscle aches; Skin: Sweating, tingling.

The sudden cessation of use of alcohol or tranquilizers can cause seizures, strokes, or heart attacks in high risk patients. A medically supervised detox can minimise an individual's symptoms of withdrawal and decrease the risk of possible complications. Some of the potentially hazardous symptoms of alcohol and tranquillizer withdrawal are: Grand mal seizures; Heart attacks; Strokes; Delirium tremens, Hallucination.(1);

- 4. Evidence of tolerance;
- 5. Progressive neglect of alternative pleasures or interests because of substance use;
- 6. Persisting with use despite clear evidence of overtly harmful consequences

Skinner and Allen (1982) found that clinicians treating patients with Alcohol

Dependence often find that their patients report symptoms and signs that are very different from what the textbooks describe.

Despite this, certain elements have been grouped as essential in ADS. These include:

- Narrowing in the repertoire (internal and external cues to drink) of drinking behaviour
- Salience of drink-seeking behaviour
- Increased tolerance to alcohol
- o Repeated withdrawal symptoms
- Repeated relief from/avoidance of withdrawal symptoms by drinking
- o A subjective awareness of a compulsion to drink
- o Relapse of the syndrome after a period of abstinence

Moreover, these elements vary in the degree to which they are present or experienced, and thus the syndrome has a *range of severity*. Further, they characterise dimensions along which clinicians can organise the information obtained from the patient (2).

#### Craving

Craving is "aversive, confusing, intrusive, frustrating, and exasperating". It can control thoughts and tends to keep people awake at night, even causing irrational words and actions from people who might otherwise be reasonable.

A number of addiction theorists hypothesise that *craving* plays an important role in both acquisition and maintenance of dependence on a drug, like alcohol.

Tiffany and Conklin (2000) theorised that craving has two prominent features:

- 1. It tends to be highly situational i.e. specifically and easily triggered by stimuli that have earlier association with use of alcohol.
- 2. Its experience can persist beyond the point of abstinence/cessation of drinking. (3)

#### **Coping with Craving**

Since craving has been described as aversive, an obvious corollary is that individuals who experience craving will find some ways to *cope* with the craving.

Coping refers to "behaviour that protects people from being harmed by problematic [social] experience". It consists of behaviour(s) that mediate the impact of issues like alcohol withdrawal, stress, societal restrictions, aggression, etc. on individuals.

Pearlin and Schooler (1978) theorise that coping behaviour(s) perform their protective functions in one of three possible ways –

- 1. Removing or changing conditions that give rise to the problem
- 2. "Perceptually controlling the meaning" of an experience in a way that neutralises or diffuses the aspect of the experience that is problematic.
- 3. Ensuring that the emotional consequences of the problem are kept within "manageable bounds". (4)

According to Fryndenberg & Lewis (2011), coping strategies can be both Productive and Unproductive.

Productive Coping Strategies – These entail dealing with the problem, and finding
ways to protect self from the psychologically damaging consequences of a particular
emotion/situation/event, while simultaneously making the attempt "to remain
physically active and socially connected".

Some examples include seeking social support, focussing on solving the problem, relaxation techniques, physical recreational activities like sports, relaxing diversions like art and dance, acceptance, and seeking professional help.

 Negative Coping Strategies – These generally encompass the use of avoidance strategies. These are usually associated with reduced ability or lack of ability to cope with stressors. Some examples include worrying, wishful thinking, ignoring the problem, withdrawing from social circle, self-blame, and acting out. (5)

#### **Jacobsen's Progressive Muscle Relaxation (JPMR)**

"An anxious mind cannot exist in a relaxed body". This quote by Dr Edmund Jacobson, is the basis for JPMR. (6)

It is the therapeutic technique of choice for use in stress and anxiety management.

JPMR was created such that it would eventually be something that the practitioner [i.e. patient] would be able to automatically and unconsciously monitor and release unwanted tension.

The technique includes the "Tension–Release" cycle (e.g. make a tight fist and then release) which has been combined with a focus on breathing. It is aimed at getting in touch with the individual's tension and the body's response, and then letting it go in a controlled manner.

Freeman (2001) suggests that PMR and other muscle-based relaxation variations convey health benefits in three ways:

- 1. Utilizing the effects of PMR to manipulate autonomic responses
- 2. Increases or activates the production of opiates
- 3. Promotes optimal immune function

The PMR method - strong record of clinical efficacy, acknowledged as standard strategy for a number of somatic states, including anxiety and stress. (7)

#### Music

Music is a "dynamic medium" that is used for inspiration, and relaxation, often on a daily basis, by many people. With this as the basis, music now plays a larger role in health and healing. Music therapy or music-based interventions are an alternative treatment route

focussed on helping patients deal with physical, emotional, and cognitive problems. It aims to enhance social or interpersonal, affective, cognitive, and behavioural functioning.

Research also shows that music is also effective at reducing muscle tension and anxiety and promotes relaxation, verbalisation, group cohesiveness and interpersonal relationships (8)

In the theory of music literature, the core assumption is on the *functions* of music. Music is generally composed or played for emotional expression. It is used to contain behaviours, and trigger cognitions. A 2007 study with adolescents found that apart from entertainment, healthy individuals used music to relax, distract themselves from certain emotions, or even to discharge these emotions, energise themselves, offer comfort or solace. Music is found to provoke sensory images within individuals - the strength of which differs from person to person.

Music also works in enabling people to sense, recognise, and express inner physical, psychological, emotional, or cognitive motions that play a role in their daily lives.

The creation of music leads to expression and containment of the emotions at the same time.

This is termed the *containing power of music*.

Society often frowns upon the expression of certain emotions like anger through aggression. Music has the power to let people experience emotion and express it without acting on it in reality.

Thus, music therapy works by applying the containing power of music and its psychobio-social aspects in a systematic manner to influence people (9)

Studies have demonstrated neurological pathways that imply application of music therapy in individuals with substance abuse problems, since, music stimulates brain processes that affect the production of certain endorphins in receptors (DRD2). The long-term use of substances severely impairs and/or damages these pathways. (8)

In a 2001 study by Daveson and Edwards, female inmates in jail reported that felt more relaxed, less stressed, and could express themselves better after 12 music therapy sessions. Patients also indicate reduction in anger, stress and frustration. Thus, research has indicated that music therapy or music-based interventions can help to move coping skills from *mainly aggressive* behaviour to *general behaviour* (10)

#### **Review of Literature**

#### **Alcohol and Stress**

(In the literature, stress is used as an umbrella term for anxiety, tension, stress, defensiveness, and associated feelings.)

Fox et al (2007) conducted a study with 20 treatment seeking ADS patients using guided imagery to imagine a "recent personal stressor, personal alcohol cue-related stressor, and a neutral imagery situation" over 3 sessions, one per session in random order. Exposure to stress and to alcohol cues each produced significant increases in alcohol craving, anxiety, and negative emotions and decreases in positive emotions.

Stress-induced alcohol craving was significantly correlated with increases in sadness, anger, and anxiety ratings, but alcohol cue-induced craving was associated with decreases in positive affect (joy and neutral relaxed state) and increases in anxiety and fear ratings. (11)

Duka et al. (2006) found in patients with multiple episodes of withdrawals from alcohol, associated craving, and anxiety. (12)

In a similar study conducted in 2000 by Sinha et al., it was observed that there were significant increases in the level of cocaine and alcohol craving with stress and drug cues imagery but not with neutral-relaxing imagery.

They also found that similar increases in subjective anxiety, heart rate and salivary cortisol levels are produced by stress and drug cues.

It was also found that there are significant increases in ratings for negative emotions and decreases in ratings for positive emotion for stress and drug cue conditions as compared to the neutral condition. (13)

#### Alcohol, Stress, and Relapse

In the 2004 meeting of the Research Society on Alcoholic Meeting Symposium, Sinha presented clinical evidence that increased sensitivity to craving increases risk for relapse; stress can cause anxiety like symptoms through craving; and that there is sufficient evidence to conclude that stress is involved in a relapse. (14)

Sinha and Li (2006) found that major factors contributing to high rates of relapse are stress and drug related cues. Further, there is an overlap in the brain areas that process stress and drug cue-induced craving, including in the medial prefrontal cortex, anterior and posterior cingulate cortex, striatal and postular insula regions; and these regions have been associated with craving state and increased susceptibility to relapse. (15)

#### **Craving and Stress**

Gruser, Morsen and Flor (2006) conducted a study on the level of craving in 50 problem drinkers, and occasional drinkers. The problem drinkers were found to have higher amount of craving accompanied by increased stress-distress; along with a higher tendency to use inadequate (negative) coping strategies.

Further, craving was found to be a significant predictor of craving. They concluded that there needs to be a focus on alternative coping strategies that would be beneficial in the management of craving. (16)

Dharmadhikari and Sinha (2015) described craving as the *psychic pain of addiction*, and that it was the *obstacle* to abstinence. Craving is what turns drug-taking behaviour into compulsive drug-taking behaviour. (17)

Swift and Stout (1992) found that craving and anxiety stress share many similar attributes, including comparable response to pharmacological agents. In their work with 32

patients who used opioids, they found the highest positive correlation between anxiety and craving. (18)

#### **Coping with Stress and Use of Music**

Labbe et al. (2007) hypothesised that listening to relaxing classical music after being exposed to a stressor should result in "significant reductions in anxiety, anger, and sympathetic nervous system arousal, and increased relaxation compared to those who sit in silence or listen to heavy metal music". Their results indicated that listening to classical music, after exposure to a stressor, significantly reduces negative emotional states and physiological arousal compared to listening to heavy metal music or sitting in silence. (19)

A meta-analysis of 22 studies by Pelletier (2004), showed that arousal due to stress is significantly reduced with music and music assisted relaxation techniques. Stress, including anxiety, fear, and tension, was found to significantly influenced by music, and strong positive correlations were observed with increased relaxation and the playing of music.

The strongest correlations were found with classical, instrumental music without lyrics, and with regular, rhythmic patterns, and no extreme changes (e.g. a beat drop). (20)

In a 2001 study by Knight and Rickard, they exposed 87 participants to a cognitive stressor task, either in presence of classical, instrumental music, or in silence. When the two groups were compared on physiological and subjective (psychological) measures of anxiety, it was found that exposure to music prevented stress induced stress induced physical arousal, and thus music acts as an effective anxiolytic. (21)

#### **Alcohol and Music**

Silverman found significant difference in the readiness to change alcohol-use behaviours between patients who were given music-based interventions and verbal therapy.

Though not significant, the patients in the music group were also found to have lower craving scores. (22)

#### Stress and PMR

In 2015, Kaur and Kaur found that PMR was effective in reducing stress levels of patients admitted for alcohol deaddiction, significant at 0.05 level. (23)

In her 2014 study with staff nurses in Vadodara, Patel found significant reduction in stress levels experienced by nurses with the use of Progressive Muscle Relaxation through pre- and post-test measures. (24)

Bommareddi et al. (2014) conducted a study with 30 patients who are living with HIV, 13% of whom had abnormal anxiety, and the rest has the increased stress levels associated with living with HIV. Comparing pre- and post-test measures of stress with the use of PMR, the reduction in stress levels was found to be significant at 0.001 level. (25)

#### Rationale of the Study

Music is an adaptive, emotion-based coping strategy, and research has shown that music-based interventions have a positive effect on levels of stress, aggression, and frustrations. Since these emotions are also associated with craving, this study aims to find if music will work in a similar manner to help patients deal with craving for alcohol.

The control technique of JPMR is selected based on research evidence that indicates its benefit with the management of stress, anxiety, depression, aggression, and frustration.

#### **Need for the Study**

As seen through the review of literature, alcohol craving and stress and correlated with relapse. Further, the use of music has demonstrated significant reduction in the level of stress experienced across various clinical and non-clinical populations.

#### **GAP IN THE KNOWLEDGE**

Though there are studies on use of music to cope with cocaine withdrawal, there is no study conducted, especially in the Indian scenario, on the effect of music on coping with craving alcohol.

If the effect is found to be significant, it can create an avenue for further research, and provide a simple, cost-free addition to treatment of patients with ADS.

#### Methodology

#### Aim

To compare the effectiveness of music and progressive muscle relaxation on craving alcohol and perceived ability to cope with craving in patients with alcohol dependence syndrome.

## **Objectives**

- To compare the pre and post-test measures of craving and coping for the two groups (within groups).
- To check the difference in the pre and post-test measures of craving and coping in the two groups (between groups).
- 3. To analyse the responses obtained through a Single Question Exit Interview, to understand patients' subjective perception about the music and the muscle relaxation

#### **Hypothesis**

- There is no difference in the effectiveness of music and progressive muscle relaxation on craving alcohol
- 2. There is no difference in the effectiveness of music and progressive muscle relaxation on perceived ability to cope with craving alcohol.

#### Sampling

- Size -10 patients in each group, so a total of 20 patients will be selected.
- Method Purposive sampling will be used.

- Design Randomized parallel intervention trial
- Criteria
  - Inclusion criteria
    - Patients with ADS
    - Adults in the age range of 18-60, of either gender
    - Abstinent for at least 1 week
  - o Exclusion criteria
    - Any other known psychiatric disorder/severe medical condition
    - Use/abuse of substances other than alcohol and nicotine
    - At risk for self-harm or suicide
  - o Drop-out criteria
    - Less than 75% compliance
    - Relapse (defined as a return to drinking behaviour)

The study duration will be 1 year, conducted on patients from Mangalore.

#### Tools to be used in the study

Three scales will be used in the study, along with a single question exit interview. Further, recorded versions of music and PMR will be used to ensure uniformity in delivery of the intervention.

#### 1. URICA Scale

The University of Rhode Island Change Assessment (URICA) Scale is designed to assess the change readiness of an individual. It acts as a screening tool for assessment of the stage of change a patient with ADS is at, based on Prochaska's Transtheoretical Model of Change.

The scale has been found to have excellent reliability and was a significant predictor of

treatment dropout and retention. The scale also showed moderate reliability as a predictor of patient prognosis. (26,27)

#### 2. Alcohol Urge Questionnaire (AUQ)

The AUQ is a self-report measure of craving alcohol, with eight items, with high internal consistency (0.91); and high test-retest reliability of 0.82 after 24 hours; as well as suitable construct validity. (28)

#### 3. Visual Analogue Scale (VAS)

The VAS is a line 100mm in length, with both the ends indicating extremes of the construct being assessed. Used generally to assess pain, VAS measures have been found to be reliable and valid measures of a number of constructs as needed. The VAS used here ranges from Completely Unable to Cope and Completely Able to Cope. The patient will indicate their subjective perception of their own ability to cope with craving alcohol.

#### 4. Single Question Exit Interview (SQI)

Each patient will be asked a single question during the final debriefing on the last day of the study. The question will be "Please describe your experience with the music/exercise". Their answers will be recorded verbatim and will be translated from Kannada as needed.

#### 5. The music

Based on the reviewed literature, Raga Bhairavi and Ahir Bhairav, played on the flute with no lyrics sung will be used in the study. (20,29–31)

The music will be played to the patients through a speaker, keeping the volume constant across all patients.

#### 6. The Progressive Muscle Relaxation

A twenty-minute PMR based on Jacobsen's Progressive Muscle Relaxation was developed and will be recorded in English and Kannada. (32) This will be done to ensure uniformity of delivery of instructions across patients.

#### Procedure

Ethical approval will be sought from the Institutional Committee. Permission will be sought from the head of the rehabilitation facility, as well as from the treating psychiatrist for each individual patient. Patients will be recruited at random from the rehabilitation centre.

After an intake interview to ensure that they meet the required criteria and providing them with all the information regarding the study, informed consent will be attained. They will be allocated to either the music group or PMR group randomly through a sequence generated through the randomizer..

Then, the URICA will be administered to obtain baseline motivation levels on Day 1, followed by AUQ, VAS for Coping. Then the first session of the assigned intervention will be conducted. On subsequent days, further sessions of the intervention will be conducted.

AUQ and VAS measurements will be taken on Day 3 and Day 5.

Music will be played at a constant volume across days and patients, and the PMR sessions will carried out as described above. On the final day, patients will be debriefed about the study and the SQI will be conducted.



Figure 1: The Process of the Study

#### **Analysis of Data**

Data will be analysed using student paired t test (pre- and post-test measures), and student unpaired t test (between post-test measures of study and control group.

Statistical package for social sciences (SPSS) software version 17.0 will be used for analysis of the data.

#### **Ethical considerations**

Ethical considerations of consent, confidentiality, competence, and non-maleficence will be adhered to in the strictest of manner

## **Implications**

This study will provide additional information towards reducing relapse in ADS patients.

This study could provide an easily available, user-friendly tool for reducing relapse in ADS patients. This study will add information to the existing pool of literature on coping, craving, alcohol dependence, and music as a coping strategy.

#### References

- Drug and Alcohol Withdrawal Symptoms Addictions and Recovery [Internet]. [cited
   2020 Apr 15]. Available from: https://www.addictionsandrecovery.org/withdrawal.htm
- Skinner HA, Allen BA. Alcohol dependence syndrome: Measurement and validation. J Abnorm Psychol [Internet]. 1982 [cited 2020 Jan 10];91(3):199–209. Available from: http://doi.apa.org/getdoi.cfm?doi=10.1037/0021-843X.91.3.199
- 3. Tiffany ST, Conklin CA. A cognitive processing model of alcohol craving and compulsive alcohol use. Addiction. 2000 Aug 10;95(8):145–53.
- 4. Pearlin LI, Schooler C. The structure of coping. J Health Soc Behav. 1978;19(1):2–21.
- 5. Frydenberg E, Lewis R. Boys play sport and girls turn to others: Age, gender and ethnicity as determinants of coping. J Adolesc. 1993;16(3):253–66.
- 6. Jacobson E. Progressive Relaxation. Am J Psychol. 1987;100(3/4):522.
- 7. Mackereth PA, Tomlinson L. therapists and patients [Internet]. Progressive Muscle Relaxation A Remarkable Tool For Therapists And Patients. Elsevier Ltd; 2010 [cited 2020 Jan 12]. 82 p. Available from: http://dx.doi.org/10.1016/B978-0-7020-3082-6.00008-3
- 8. AMTA. Definition and Quotes about Music Therapy | Definition and Quotes about Music Therapy | American Music Therapy Association (AMTA) [Internet]. 2017 [cited 2020 Jan 12]. Available from: https://www.musictherapy.org/about/quotes/
- 9. Hakvoort L, Bogaerts S, Thaut MH, Spreen M. Influence of music therapy on coping skills and anger management in forensic psychiatric patients: An exploratory study. Int J Offender Ther Comp Criminol. 2015 Jul 19;59(8):810–36.

- 10. Daveson BA, Edwards J. A descriptive study exploring the role of music therapy in prisons. Arts Psychother [Internet]. 2001 May [cited 2020 Jan 12];28(2):137–41.
  Available from: https://linkinghub.elsevier.com/retrieve/pii/S0197455600000897
- 11. Sinha R, Fox HC, Hong KIA, Hansen J, Tuit K, Kreek MJ. Effects of adrenal sensitivity, stress- and cue-induced craving, and anxiety on subsequent alcohol relapse and treatment outcomes. Arch Gen Psychiatry. 2011 Sep 5;68(9):942–52.
- 12. Duka T, Townshend JM, Collier K, Stephens DN. Kindling of withdrawal: A study of craving and anxiety after multiple detoxifications in alcoholic inpatients. Alcohol Clin Exp Res. 2002;26(6):785–95.
- 13. Sinha R, Fuse T, Aubin LR, O'Malley SS. Psychological stress, drug-related cues and cocaine craving. Psychopharmacology (Berl). 2000;152(2):140–8.
- 14. Breese GR, Chu K, Dayas C V., Funk D, Knapp DJ, Koob GF, et al. Stress enhancement of craving during sobriety: A risk for relapse. In: Alcoholism: Clinical and Experimental Research. 2005. p. 185–95.
- Sinha R, Li CSR. Imaging stress- and cue-induced drug and alcohol craving:
   Association with relapse and clinical implications. Vol. 26, Drug and Alcohol Review.
   2007. p. 25–31.
- 16. Grüsser SM, Mörsen CP, Wölfling K, Flor H. The relationship of stress, coping, effect expectancies and craving. Eur Addict Res. 2006 Dec;13(1):31–8.
- 17. Sinha VK D. Psychological Management of Craving. J Addict Res Ther. 2015;06(02).
- 18. Swift RM, Stout RL. The relationship between craving, anxiety, and other symptoms in opioid withdrawal. J Subst Abuse [Internet]. 1992 [cited 2020 Jan 12];4(1):19–26. Available from: http://www.ncbi.nlm.nih.gov/pubmed/1320971

- Labbé E, Schmidt N, Babin J, Pharr M. Coping with stress: The effectiveness of different types of music. Appl Psychophysiol Biofeedback. 2007 Dec;32(3-4):163-8.
- Pelletier CL. The effect of music on decreasing arousal due to stress: A meta-analysis.
   Vol. 41, Journal of Music Therapy. American Music Therapy Association; 2004. p.
   192–214.
- Knight WEJ, Rickard NS. Relaxing Music Prevents Stress-Induced Increases in Subjective Anxiety, Systolic Blood Pressure, and Heart Rate in Healthy Males and Females. J Music Ther. 2001;38(4):254–72.
- 22. DiClemente CC, Hughes SO. Stages of change profiles in outpatient alcoholism treatment. J Subst Abuse. 1990;2(2):217–35.
- 23. Sharma V, Kaur S. Spiritual wellness among aggressive adolescents: Efficacy of Raga Bhairavi. Psychomusicology Music Mind, Brain. 2017 Dec;27(4):350–4.
- 24. Patel MP. "A Study to Assess the Effectiveness Of Progressive Muscle Relaxation Therapy on Stress among Staff Nurses Working In Selected Hospitals at Vadodara City" [Internet]. Vol. 3. [cited 2020 Jan 12]. Available from: www.iosrjournals.orgwww.iosrjournals.org
- 25. Bommareddi P, Prabha Valsaraj B, Bommareddi R. JACOBSON'S PROGRESSIVE MUSCLE RELAXATION (JPMR) TRAINING TO REDUCE ANXIETY AND DEPRESSION AMONG PEOPLE LIVING WITH HIV 1 2 3.
- 26. Dozois DJA, Westra HA, Collins KA, Fung TS, Garry JKF. Stages of change in anxiety: Psychometric properties of the University of Rhode Island Change Assessment (URICA) scale. Behav Res Ther. 2004 Jun;42(6):711–29.
- 27. Hasler G, Klaghofer R, Buddeberg C. The University of Rhode Island Change

- Assessment Scale (URICA) Psychometric Testing of a German Version. PPmP Psychother Psychosom Medizinische Psychol [Internet]. 2003 Sep [cited 2020 Jan 28];53(9–10):406–11. Available from: http://www.thiemeconnect.de/DOI/DOI?10.1055/s-2003-42172
- 28. Drobes DJ, Thomas SE. Assessing craving for alcohol. Alcohol Res Heal J Natl Inst Alcohol Abus Alcohol [Internet]. 1999;23(3):179–86. Available from: http://www.ncbi.nlm.nih.gov/pubmed/10890813
- 29. Kotwal MR, Rinchhen CZ, Ringe V V. Stress reduction through listening to Indian classical music during gastroscopy. Diagn Ther Endosc [Internet]. 1998 [cited 2020 Feb 15];4(4):191–7. Available from: http://www.ncbi.nlm.nih.gov/pubmed/18493472
- 30. PV BD. Stress Reduction Through Listening Indian Classical Music. Innovare J Heal Sci. 2014;2(2):4–8.
- 31. Scherer KR. Which Emotions Can be Induced by Music? What Are the Underlying Mechanisms? And How Can We Measure Them? J New Music Res [Internet]. 2004 Sep [cited 2018 Nov 18];33(3):239–51. Available from: http://www.tandfonline.com/doi/abs/10.1080/0929821042000317822
- 32. Mushtaq B, Khan AA. Jacobson Muscle Relaxatation Technique (Jpmr) (20 Min) JOJ Nurse Health Care. JOJ Nurse Heal Care [Internet]. 2018 [cited 2020 Jan 12];8(1). Available from: https://juniperpublishers.com/online-submission.php

## **Appendix**

- 1. Client Information Sheet/Informed Consent Form
- 2. URICA Scale
- 3. AUQ
- 4. VAS for Coping
- 5. Patient Register
- 6. Record Sheet
- 7. Randomised list of assigning conditions
- 8. Permissions for
  - a. URICA
  - b. AUQ
- 9. Letter of permission from treating psychiatrist

#### 1. Client Information Sheet/Informed Consent Form



#### KASTURBA MEDICAL COLLEGE, MANGALORE

#### DEPARTMENT OF PSYCHIATRY

#### SUBJECT INFORMATION SHEET

Study: Comparison Between the Use of Music and Relaxation Training on Craving Alcohol in Patients with Alcohol Dependence Syndrome: A Pilot Study

Investigator: Shradha Chandrasekar, student, MSc Clinical Psychology, KMC Mangalore.

Guide: Dr Keshava Pai, Professor and Head, Dept. of Psychiatry, KMC Mangalore.

#### STUDY AND INVESTIGATORS

This study involves comparison between two techniques to see which works better to help cope with alcohol craving. One of the techniques is music, the other is a relaxation technique called Progressive Muscle Relaxation.

It is being conducted by Shradha Chandrasekar, student, pursuing MSc Clinical Psychology at Kasturba Medical College, Mangalore, under the guidance of Dr Keshava Pai, professor and Head of Department of Psychiatry at Kasturba Medical College, Mangalore.

Your participation in this study is wholly voluntary, and you should only agree to it after reading the following information and clarifying any queries you may have.

#### PROCEDURE OF THE STUDY

If you agree to participate in this study, you will be assigned either of the two techniques randomly. You will be explained how the technique assigned to you is to be used. Your urge to drink and how well you think you can cope with it will be assessed on this first day.

At three days, and then again at five days, your craving and coping again be assessed.

#### BENEFIT OF THE STUDY

When the techniques are found to be useful, they can be used as an additional treatment tool in therapy of patients with alcohol dependence.

#### SAFETY INFORMATION

Both techniques are non-invasive and will not produce any side-effects.

#### RISKS AND DISCOMFORT

However, if at any point during the study you feel uncomfortable, you can contact the Investigator (cshradha1@gmail.com) or the Guide (paikeshava@gmail.com) through email or on the KMC Attavar OPD office number 0824 2445858, Extn – 5335, or by asking the operator for Psychiatry OPD.

#### WITHDRAWAL FROM THE STUDY

You can withdraw from the study at any point without your medical care or legal rights being affected.

The Investigator or Guide may terminate your participation in the study at any point if such a situation may arise.

#### CONFIDENTIALITY

All information collected from you will be kept confidential. If the data are used for publication in psychological journals, no identifying information of any kind will be used with your permission.

If you agree to participate in the study the Ethics Committee and the regulatory authorities will not need your permission to look at your health records both in respect of the current study and any further research that may be conducted in relation to it, even if I withdraw from the trial.

#### **FURTHER INFORMATION**

You may ask any question or clarification or extra information at any point from the Investigator or the Guide, and they will be available to answer your questions and concerns. You will be given a copy of this sheet and of the Informed consent form for your records.



#### KASTURBA MEDICAL COLLEGE, MANGALORE

#### DEPARTMENT OF PSYCHIATRY

#### **INFORMED CONSENT FORM**

#### **SUBJECT COPY**

| Subject's Name: | Subject's Initials: |
|-------------------------|---------------------|
| Date of Birth:// | Age: |
| Mobile number: Subject: | Caregiver: |

Study: Comparison Between the Use of Music and Relaxation Training on Craving Alcohol in Patients with Alcohol Dependence Syndrome: A Pilot Study

Investigator: Shradha Chandrasekar, student, MSc Clinical Psychology, KMC Mangalore.

Guide: Dr Keshava Pai, Professor and Head, Dept. of Psychiatry, KMC Mangalore.

I have read/I have been explained the study and I confirm that I have understood the information sheet for the study. I also understand that I can contact the Investigator or the Guide at any point through email for further clarification/information.

MUSIC AND JPMR WITH ADS: A PILOT STUDY

I understand that my participation in the study is voluntary and that I am free to

withdraw at any time, without giving any reason, without my medical care or legal rights

being affected.

I also understand that the Investigator or Guide may terminate my participation in the

study at any point if such a situation may arise.

I understand that the Ethics Committee and the regulatory authorities will not need

my permission to look at my health records both in respect of the current study and any

further research that may be conducted in relation to it, even if I withdraw from the trial.

However, I understand that my identity will not be revealed in any information

released to third parties or published. I agree not to restrict the use of any data or results that

arise from this study provided such a use is only for scientific purpose(s).

Signature/Thumb Impression of

Signature of Investigator with date

Subject/Legal Representatives with date

Contact details: Investigator: Shradha Chandrasekar

cshradha1@gmail.com

Guide: Dr Keshava Pai

paikeshava@gmail.com

Office number: 0824 - 2445858, Extn – 5335

29



## KASTURBA MEDICAL COLLEGE, MANGALORE DEPARTMENT OF PSYCHIATRY

#### INFORMED CONSENT FORM

#### **INVESTIGATOR COPY**

| Subject's Name: | Subject's Initials: |
|-------------------------|---------------------|
| Date of Birth:/ | Age: |
| Mobile number: Subject: | Caregiver: |

Study: Comparison Between the Use of Music and Relaxation Training on Craving Alcohol in Patients with Alcohol Dependence Syndrome: A Pilot Study

Investigator: Shradha Chandrasekar, student, MSc Clinical Psychology, KMC Mangalore.

Guide: Dr Keshava Pai, Professor and Head, Dept. of Psychiatry, KMC Mangalore.

I have read/I have been explained the study and I confirm that I have understood the information sheet for the study. I also understand that I can contact the Investigator or the Guide at any point through email for further clarification/information.

MUSIC AND JPMR WITH ADS: A PILOT STUDY

I understand that my participation in the study is voluntary and that I am free to

withdraw at any time, without giving any reason, without my medical care or legal rights

being affected.

I also understand that the Investigator or Guide may terminate my participation in the

study at any point if such a situation may arise.

I understand that the Ethics Committee and the regulatory authorities will not need

my permission to look at my health records both in respect of the current study and any

further research that may be conducted in relation to it, even if I withdraw from the trial.

However, I understand that my identity will not be revealed in any information

released to third parties or published. I agree not to restrict the use of any data or results that

arise from this study provided such a use is only for scientific purpose(s).

Signature/Thumb Impression of

Signature of Investigator with date

Subject/Legal Representatives with date

Contact details: Investigator: Shradha Chandrasekar

cshradha1@gmail.com

Guide: Dr Keshava Pai

paikeshava@gmail.com

Office number: 0824 - 2445858, Extn – 5335

31



## ಕಸ್ಕೂರ್ಬಾ ಮೆಡಿಕಲ್ಕಾಲೇಜು, ಮಂಗಳೂರು

## ಮನೋರೋಗಚಿಕಿತ್ತಾ ಇಲಾಖೆ

## ವಿಷಯದ ಮಾಹಿತಿ ಪತ್ರ

## ಶೀರ್ಷಿಕೆ :

ಮಧ್ಯಪಾನಅವಲಂಚಿತ ಸಿಂಡ್ರೋಮ್ ಇರುವ ರೋಗಿಗಳಲ್ಲ ಮಧ್ಯಪಾನದ ಚಟಜಡಿಸುವುದಕ್ಕೆ ಸಂಗೀತ ಮತ್ತು ವಿಶ್ರಾಂತಿ ತರಭೇತಿಯ ನಡುವಿನ ಹೋಲಕೆಯ ಅಧ್ಯಯನ. ಇದುತನಿಖೆದಾರರ ಅಧ್ಯಯನ.

<u>ತನಿಖಾಧಿಕಾರಿ :ಶ್ರದ್ಧಾಚಂದ್ರಶೇಖರ್, MSc ಮನಃಶಾಸ್ತ್ರ ವಿದ್ಯಾರ್ಥಿ, ಕೆ.ಎಂ.ಸಿ ಮಂಗಳೂರು</u>

<u>ಮಾರ್ಗದರ್ಶಕರು</u>:ಡಾ। ಕೇಶವ ಪೈ, ಪ್ರಾಧ್ಯಾಪಕ ಮತ್ತು ಮುಖ್ಯಸ್ಥ,ಮನೋರೋಗಚಿಕಿತ್ಸಾ ವಿಭಾಗ ಕೆ.ಎಂ.ಸಿ ಮಂಗಳೂರು

## ಅಧ್ಯಯನ ಮತ್ತುತನಿಖೆದಾರರು :

ಈ ಅಧ್ಯಯನವು ಮದ್ಯಸಾರ ಪಾನೀಯ ಸೇವಿಸುವ ರೋಗಿಗಳ ಕಡುಬಯಕೆಯನ್ನು ನಿಭಾಯಿಸಲು ಸಹಾಯ ಮಾಡುವಎರಡು ತಂತ್ರಗಳ ನಡುವಿನ ಹೋಅಕೆಯಾಗಿದೆ.ತಂತ್ರಗಳಲ್ಲ ಒಂದು ಸಂಗೀತವೆಂದರೆ, ಇತರ ಪ್ರಗತಿಶೀಲ ಸ್ವಾಯುವಿನ ವಿಶ್ರಾಂತಿತಂತ್ರವಾಗಿದೆ.

ಈ ಅಧ್ಯಯನವನ್ನು ಮಂಗಳೂಲಿನ ಕಸ್ತೂರ್ಬಾ ಮೆಡಿಕಲ್ಕಾಲೀಜನಲ್ಲಿ MSC ಮನಃಶಾಸ್ತ್ರ ವ್ಯಾಸಂಗ ಮಾಡುತ್ತಿರುವವಿದ್ಯಾರ್ಥಿ, ಶ್ರದ್ಧಚಂದ್ರಶೇಖರ್ಇವರುಡಾ ಕೇಶವ ಪೈ, ಪ್ರಾಧ್ಯಾಪಕ ಮತ್ತು ಮುಖ್ಯಸ್ಥ, ಮನೋರೋಗಚಿಕಿತ್ಸಾ ವಿಭಾಗ ಕೆ.ಎಂ.ಸಿ ಮಂಗಳೂರು ಇವರ ಮಾರ್ಗದರ್ಶನದಲ್ಲ ನಡೆಸಲಾಗುತ್ತದೆ. ನನ್ನ ಪಾಲ್ಗೊಳ್ಳುವಿಕೆಯು ಸ್ವಯಂಪ್ರೇರಿತವಾಗಿರುವುದನ್ನು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ. ಕೆಳಗಿನ ಮಾಹಿತಿಗಳನ್ನು ಓದಿದ ನಂತರ ನೀವು ಅದನ್ನು ಒಪ್ಪಿಕೊಳ್ಳಬೇಕು.ನಿಮ್ಮಯಾವುದೇ ಪ್ರಶ್ನೆಯನ್ನುಇಲ್ಲಸ್ಪಷ್ಠೀಕರಿಸಬಹುದು.

## ಅಧ್ಯಯನದಕಾರ್ಯವಿಧಾನ :

ಈ ಅಧ್ಯಯನದಲ್ಲ ಪಾಲ್ಗೊಳ್ಳಲು ನೀವು ಒಪ್ಪಿಕೊಂಡರೆ, ನೀವು ಗೊತ್ತಿಲ್ಲದಎರಡು ತಂತ್ರಗಳನ್ನು ನಿಯೋಜಸಬೇಕಾಗುತ್ತದೆ.ನಿಮಗೆ ನಿಯೋಜಸಲಾದತಂತ್ರವನ್ನು ಹೇಗೆ ಬಳಸಬೇಕು ಎಂದು ಈ ಅಧ್ಯಯನದಲ್ಲ ವಿವರಿಸಲಾಗುತ್ತದೆ.ಕುಡಿಯಲು ನಿಮ್ಮ ಪ್ರಜೋದನೆ ಮತ್ತು ನೀವು ಅ ಮೊದಲ ದಿನದಂದು ಮೌಲ್ಯಮಾಪನ ಮಾಡುವ ನಿಟ್ಟನಲ್ಲ ನೀವು ಎಷ್ಟು ಚೆನ್ನಾಗಿಯೋಚಿಸಬಹುದುಎಂದು ಈ ಅಧ್ಯಯನದಲ್ಲ ನಿರ್ಧರಿಸಲಾಗುತ್ತದೆ.

ಮೂರು ದಿನಗಳಲ್ಲ, ನಂತರ ಮತ್ತೆಐದು ದಿನಗಳಲ್ಲ, ನಿಮ್ಮಕಡುಬಯಕೆಯನ್ನು ನಿಭಾಯಿಸಲು ಮತ್ತೆ ಮೌಲ್ಯಮಾಪನ ಮಾಡಲಾಗುತ್ತದೆ.

## ಅಧ್ಯಯನದ ಪ್ರಯೋಜನಗಳು :

ಈ ಅಧ್ಯಯನದ ತಂತ್ರಗಳು ಉಪಯುಕ್ತವೆನಿಸಿದಾಗ, ಮಧ್ಯಸಾರ ಪಾನೀಯ ಸೇವಿಸುವ ರೋಗಿಗಳ ಚಿಕಿತ್ಸೆಯಲ್ಲ ಹೆಚ್ಚುವರಿ ಸಾಧನವಾಗಿ ಈ ಅಧ್ಯಯನವನ್ನು ಬಳಸಬಹುದಾಗಿದೆ.

## ಸುರಕ್ಷತೆಯ ಮಾಹಿತಿ:

ಈ ಅಧ್ಯಯನದಎರಡೂ ವಿಧಾನಗಳಲ್ಲ ಪಾಲ್ಗೊಳ್ಳುವುದರಿಂದ ಯಾವುದೇಅಪಾಯವಿರುವುದಿಲ್ಲ ಇದುಯಾವುದೇ ಅಡ್ಡಪರಿಣಾಮಗಳನ್ನು ಉಂಟುಮಾಡುವುದಿಲ್ಲ.

## <u>ಅಪಾಯ ಮತ್ತುಅಸ್ವಸ್ಥತೆ :</u>

ಈ ಅಧ್ಯಯನದಲ್ಲ ಪಾಲ್ಗೊಳ್ಳುವುದರಿಂದ ನೀವು ಅನಾನುಕೂಲತೆಯನ್ನು ಅನುಭವಿಸಿದರೆ ಅಥವಾ ಈ ಅಧ್ಯಯನದ ಬಗ್ಗೆ ಯಾವುದೇ ಮಾಹಿತಿ, ಪ್ರಶ್ನೆಗಳನ್ನು ಹೊಂದಿದ್ದರೆ, ತನಿಖಿದಾರರನ್ನು(cshradha1@gmail.com)ಅಥವಾ ಮಾರ್ಗದರ್ಶಿಯ (paikeshava@gmail.com) ಈ ಇಮೇಲ್ಐಡಿಯನ್ನು ಬಳಸಿಕೊಳ್ಳಬಹುದು. ಅಥವಾ, ಕೆ.ಎಂ.ಸಿ ಅತ್ತಾವರದOPDಅಫೀಸ್ನದೂರವಾಣಿ ಸಂಖ್ಯೆ: 0824- 2445858, - 5335, ಹಾಗೂ ಅಪರೇಟರನ್ನು ಕೇಳುವ ಮೂಲಕ ಸಂಪರ್ಕಿಸಬಹುದು.

## ಅಧ್ಯಯನದಿಂದಹಿಂತೆಗೆದುಕೊಳ್ಳುವ ಹಕ್ತು:

ಈ ಅಧ್ಯಯನದಲ್ಲನನ್ನ ವೈದ್ಯಕೀಯಆರೈಕೆಅಥವಾ ಕಾನೂನಿನ ಹಕ್ಕಿನಿಂದಯಾವುದೇ ಪರಿಣಾಮವಿಲ್ಲದೆಯೇ, ಯಾವುದೇಕಾರಣವನ್ನು ಹೇಳುವ ಮೂಲಕ ಯಾವುದೇ ಸಮಯದಲ್ಲಾದರೂ ಹಿಂಪಡೆಯಲು ನಾನು ಮುಕ್ತನಾಗಿರುತ್ತೇನೆ.

ಅಧ್ಯಯನದಿಂದ ಹಿಂತೆಗೆದುಕೊಳ್ಳುವ ಪರಿಸ್ಥಿತಿ ಉದ್ಬವವಾಗುದಾದರೆಯಾವುದೇ ಹಂತದಲ್ಲತನಿಖಾಧಿಕಾರಿಅಥವಾ ಮಾರ್ಗದರ್ಶಿಯು ನಿಮ್ಮ ಪಾಲ್ಗೊಳ್ಳುವಿಕೆಯನ್ನು ಕೊನೆಗೊಆಸಬಹುದು.

## <u>ಗೌಪ್ಯತೆ :</u>

ಈ ಅಧ್ಯಯನದಿಂದ ಒದಗಿಸಿದ ಮಾಹಿತಿಗಳನ್ನು ಗೌಪ್ಯವಾಗಿಡಲಾಗುವುದು ಮತ್ತು ವೈಜ್ಞಾನಿಕ ಪ್ರಸ್ತುತಿ ಮತ್ತುಗುರುತಿನ ಮಾಹಿತಿಯಲ್ಲದೇ ಪ್ರಕಟನೆಯರೂಪದಲ್ಲ ಮಾತ್ರ ಗುಂಪು ಡೇಟಾವನ್ನು ವರದಿ ಮಾಡಲಾಗುವುದು.ಈ ಎಲ್ಲಾಡೇಟಾವನ್ನು ಸುರಕ್ಷಿತ ಸ್ಥಳದಲ್ಲ ಇರಿಸಲಾಗುವುದು ಮತ್ತು ಈ ಸಂಶೋಧನೆಯೊಂದಿಗೆ ನೇರವಾಗಿ ತೊಡಗಿಸಿಕೊಂಡಿರುವವರಿಗೆ ಅದು ಪ್ರವೇಶವನ್ನು ಹೊಂದಿರುತ್ತದೆ.ಹಾರ್ಡ್ ಪ್ರತಿಗಳನ್ನು ಲಾಕರ್ ಒಂದು ಮತ್ತುಕೀಅಯಲ್ಲಇಡಲಾಗುವುದು.ಅದನ್ನುರಕ್ಷಕರಿಗೆಅಥವಾಅಧ್ಯಯನದಲ್ಲ ಒಳಗೊಂಡಿರುವ ಮಾರ್ಗದರ್ಶಿಗಆಗೆ ಮಾತ್ರ ಪ್ರವೇಸಿಶಬಹುದು.ಸಂಶೋಧಕರ ವೈಯಕ್ತಿಕ ಲ್ಯಾಪ್ ಚಾಪ್ ನಲ್ಲ ಮೃದುವಾದ ನಕಲು ಪತ್ರಿಗಳನ್ನು ಒಂದು ಪಾಸ್ತರ್ಡ್ನಲ್ಲ ಪೋಲ್ಡರ್ನಅ್ಲಇಡಲಾಗುವುದು.ಇದನ್ನು ಮಾತ್ರ ಸಂಶೋಧಕರುಅಥವಾ ಮಾರ್ಗದಶಕರು ಪ್ರವೇಶಿಸಬಹುದು.

## ಹೆಚ್ಚಿನ ಮಾಹಿತಿಗಾಗಿ :

ಈ ಅಧ್ಯಯನದ ಬಗ್ಗೆ ಯಾವುದೇ ಮಾಹಿತಿ, ಪ್ರಶ್ನೆಗಳನ್ನು ಹೊಂದಿದ್ದರೆ, ಅಧ್ಯಯನದಮಾರ್ಗದರ್ಶಿಯವರನ್ನು ಸಂಪರ್ಕಿಸಬಹುದು ನಿಮ್ಮ ಪ್ರಶ್ನೆ ಮತ್ತು ಕಾಳಜಗಳಗೆ ಉತ್ತರಿಸುವ ಹಕ್ಕನ್ನುಅವರು ಹೊಂದಿರುತ್ತಾರೆ. ನಿಮ್ಮಅಧ್ಯಯನದ ದಾಖಲೆಗಳ ತಿಳುವಳಕೆಯ ಮಾಹಿತಿ ಪತ್ರದ ನಕಲು ಪ್ರತಿಯನ್ನು ನಿಮಗೆ ನೀಡಲಾಗುವುದು.



## ಕಸ್ತೂರ್ಬಾ ಮೆಡಿಕಲ್ಕಾಲೇಜು, ಮಂಗಳೂರು

## ಮನೋರೋಗಚಿಕಿತ್ಸಾ ಇಲಾಖೆ

## ತಿಳುವಆಯ ಮಾಹಿತಿ ಪತ್ರ

## ತನಿ<mark>ಖೆದ್ದಾರರ ನ<del>ಕ</del>ಲು</mark>

| ವಿಷಯದ ಹೆಸರು : | | ವಿಷಯದಆರಂಭ : | |
|---|---|---|---|
| ಹುಟ್ಟದ ದಿನಾಂಕ ://_ | | ವಯಸ್ಸು : | |
| ಮೊಬೈಲ್ ಸಂಖ್ಯೆ : ವಿಷಯ : | | ಪಾಲನೆದಾರ : | _ |
| <u>ಶೀರ್ಷಿಕೆ</u> :ಮದ್ಯಪಾನಅವಲಂಜತ ಸಿಂಡ್ರೇಮ್ ಇರುವ ರೋಗಿಗಳಲ್ಲ ಮದ್ಯಪಾನದಚಟ ಜಡಿಸುವುದಕ್ಕೆ ಸಂಗೀತ<br>ಮತ್ತು ವಿಶ್ರಾಂತಿತರಭೇತಿಯ ನಡುವಿನ ಹೋಲಕೆಯಅಧ್ಯಯನ. ಇದುತನಿಖಿದಾರರಅಧ್ಯಯನ. | | | |
| <mark>ತನಿಖಾಧಿಕಾರಿ :ಶ್ರದ್ಧಾಚಂದ್ರಶೇ</mark> ಖರ್, MSc ಮನಃಶಾಸ್ತ್ರ ವಿದ್ಯಾರ್ಥಿ, ಕೆ.ಎಂ.ಸಿ ಮಂಗಳೂರು | | | |
| <mark>ಮಾರ್ಗದರ್ಶಕರು :</mark> ಡಾ। ಕೇಶವ ಪೈ, ಪ್ರಾಧ್ಯಾಪಕ ಮತ್ತು ಮುಖ್ಯಸ್ಥ, ಮನೋರೋಗಚಿಕಿತ್ಸಾ ವಿಭಾಗ ಕೆ.ಎಂ.ಸಿ<br>ಮಂಗಳೂರು | | | |
| ನಾನುಮೇಅನ | <b>ಅದ್ಯಯನದಅ</b> ಒದಗಿಸಲಾದ | ಮಾಹಿತಿಯನು | ನಾನು |

ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ.ಅಧ್ಯಯನದಉದ್ದೇಶ ಮತ್ತು ಉದ್ದೇಶಗಳು, ಅವಧಿ ಮುಗಿದ ಪರಿಣಾಮಗಳನ್ನು ನಾನು

ತಿಆಸಿಕೊಡಲಾಗಿದೆ.ನಾನು ಅಧ್ಯಯನದಬಗ್ಗೆ ಕೇ**ಳಲು ಸಮಯ ಮತ್ತು**ಅವಕಾಶವನ್ನು ಹೊಂದಿದ್ದೇನೆ. ಅಧ್ಯಯನದ

ಭಾಗವಾಗಿ

ಏನು

ಮಾಡಬೇಕೆಂದು

ನನಗೆ

ಭಾಷೆಯಲ್ಲವಿವರಿಸಲಾಗಿದೆ.ಅಧ್ಯಯನದ

ವಿವರಣೆಯನ್ನು ಸಂಪೂರ್ಣವಾಗಿ ತಿಆಸಿಕೊಡಲಾಗಿದೆ.

ವಿವರಿಸಿರುವ
ನನ್ನ ಪಾಲ್ಗೊಳ್ಳುವಿಕೆಯು ಸ್ವಯಂಪ್ರೇರಿತವಾಗಿರುವುದನ್ನು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ ಮತ್ತು ನನ್ನ ವೈದ್ಯಕೀಯಆರೈಕೆಅಥವಾ ಕಾನೂನಿನ ಹಕ್ಕಿನಿಂದಯಾವುದೇ ಪರಿಣಾಮವಿಲ್ಲದೆಯೇ, ಯಾವುದೇಕಾರಣವನ್ನು ಹೇಳುವ ಮೂಲಕ ಯಾವುದೇ ಸಮಯದಲ್ಲಾದರೂ ಹಿಂಪಡೆಯಲು ನಾನು ಮುಕ್ತನಾಗಿರುತ್ತೇನೆ.

ಅಧ್ಯಯನದಿಂದ ಹಿಂತೆಗೆದುಕೊಳ್ಳುವ ಪರಿಸ್ಥಿತಿ ಉಂಟಾಗಬಹುದಾದರೆಯಾವುದೇ ಹಂತದಲ್ಲತನಿಖಾಧಿಕಾರಿಅಥವಾ ಮಾರ್ಗದರ್ಶಿಯು ನಿಮ್ಮ ಪಾಲ್ಗೊಳ್ಳುವಿಕೆಯನ್ನು ಕೊನೆಗೊಳಸಬಹುದುಎಂದು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ.

ಈ ಅಧ್ಯಯನದಿಂದ ಒದಗಿಸಿದ ಮಾಹಿತಿಗಳನ್ನು ಗೌಪ್ಯವಾಗಿಡಲಾಗುವುದು ಮತ್ತು ವೈಜ್ಞಾನಿಕ ಪ್ರಸ್ತುತಿ ಮತ್ತುಗುರುತಿನ ಮಾಹಿತಿಯಲ್ಲದೇ ಪ್ರಕಟನೆಯರೂಪದಲ್ಲ ಮಾತ್ರ ಗುಂಪು ಡೇಟಾವನ್ನು ವರದಿ ಮಾಡಲಾಗುವುದು.ಅಧ್ಯಯನದಲ್ಲ ಭಾಗವಹಿಸುವ ನನ್ನ ನಿರ್ಧಾರ ನನ್ನಚಿಕಿತ್ಸೆಯ ಮೇಲೆ ಪರಿಣಾಮ ಜೀರುವುದಿಲ್ಲ ಎಂದು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ.

ಈ ಅಧ್ಯಯನದಉಂಟಾದ ಫಲತಾಂಶದ ಬಳಕೆಯನ್ನು ನಿಬಂಧಿಸಲು ನಾನು ಸಮ್ಮತಿಸುವುದಿಲ್ಲ ಅದನ್ನು ಸೂಕ್ತ ಅಧಿಕಾರಿಗಆಗೆ ರವಾನಿಸಬಹುದು ಮತ್ತು ಪ್ರಕಟಸಬಹುದಾಗಿದೆ.

ಅಧ್ಯಯನದಲ್ಲ ಭಾಗವಹಿಸುವ ನನ್ನ ನಿರ್ಧಾರ ನನ್ನಚಿಕಿತ್ಸೆಯ ಮೇಲೆ ಪರಿಣಾಮ ಜೀರುವುದಿಲ್ಲ ಎಂದು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ. \_\_\_\_\_

ಸಹಿ/ಹೆಬ್ಬೆರಳು ಗುರುತಿನೊಂದಿಗೆ

ತನಿಖೆದಾರರ ಸಹಿ ಮತ್ತು ದಿನಾಂಕ

ವಿಷಯ/ಕಾನೂನು ಬದ್ದಚಿತ್ರಣದ ದಿನಾಂಕ

ಸಂಪರ್ಕ ಮಾಹಿತಿ :ತನಿಖಿದಾರರು : ಶ್ರದ್ಧಾಚಂದ್ರಶೇಖರ್

cshradha1@gmail.com

ಮಾರ್ಗದರ್ಶಕರು :ಡಾ ಕೇಶವ ಪೈ

paikeshava@gmail.com

ಆಫೀಸ್ ನಂ : 0824-2445858, - 5335



# ಕಸ್ತೂರ್ಬಾ ಮೆಡಿಕಲ್ಕಾಲೇಜು, ಮಂಗಳೂರು

## ಮನೋರೋಗಚಿಕಿತ್ಸಾ ಇಲಾಖೆ

# ತಿಳುವಆಯ ಮಾಹಿತಿ ಪತ್ರ

# <u>ಬಾಗವಹಿಸುವವರ</u> ಪತ್ರ

| ವಿಷಯದ | ಹೆಸರು : | | | ವಿಷಯದಆ | ಕರಂಭ : | <b>!</b> | |
|---|---|---|---|---|---|---|---|
| ಕುಟ್ಟದ ದಿ | ನಾಂಕ :// | | | ವಯಸ್ಸು : | | | |
| ಮೊಬೈಲ್ | ಸಂಖ್ಯೆ : ವಿಷಯ : | | | ಪಾಲನೆದಾ | ರ : | | - |
| ಶೀರ್ಷಿಕ | <u>ಕೆ</u> :ಮದ್ಯಪಾನಅವಲಂಚತ<br>ಮತ್ತು ವಿಶ್ರಾಂತಿತರಭೇತೀ | | | . 0 | | · · | ೧೧೬ತ |
| <u>ತ</u> ನಿಖಾÇ | ) <del>ප</del> ಾ <b>ට</b> : | ್, MSc <b>ಮನಃಶ</b> | മുട്ട് മുന്തു കൂട്ട് കുടു | ಕೆ.ಎಂ.ಸಿ ವ | ಬಂಗಳು | ಾರು | |
| ಮಾರ್ಗ<br>ಮಂಗಳೂ | <b>ವರ್ಶಕರು :</b> ಡಾ ಕೇಶವ<br>ಾರು | ಪೈ, ಪ್ರಾಧ್ಯಾಪ <del>ಕ</del> | ಮತ್ತು ಮುಖ್ಯಸ್ಥ | ಕ್ಟ, ಮನೋ | ರೋಗಣ | ಚಿಕಿತ್ಸಾ ವಿಭಾಗ ಕ | కి.ఎం.సి |
| 7 | ಾನುಮೇಲನ | ಅಧ್ಯಯನದಲ್ಲಒ | ದೆಗಿಸಲಾದ | ವ | ර්ෂ සිට | <b>ು</b> ನ್ನು | ನಾನ |
| ಅರ್ಥಮಾ | ಡಿಕೊಂಡಿದ್ದೇನೆ.ಅಧ್ಯಯನದ | ಉದ್ದೇಶ ಮತ್ತು | ಉದ್ದೇಶಗಳು, | ಅವಧಿ ವ | ು<br>ಗಿದ | ಪರಿಣಾಮಗಳನ್ನು | ನಾನ |

ತಿಆಸಿಕೊಡಲಾಗಿದೆ.ನಾನು ಅಧ್ಯಯನದಬಗ್ಗೆ ಕೇ**ಳಲು ಸಮಯ ಮ**ತ್ತುಅವ<del>ಕ</del>ಾಶವನ್ನು ಹೊಂದಿದ್ದೇನೆ. ಅಧ್ಯಯನದ

ಭಾಗವಾಗಿ

ಏನು

ಮಾಡಬೇಕೆಂದು

ನನಗೆ

ಭಾಷೆಯಲ್ಲವಿವರಿಸಲಾಗಿದೆ.ಅಧ್ಯಯನದ

ವಿವರಣೆಯನ್ನು ಸಂಪೂರ್ಣವಾಗಿ ತಿಆಸಿಕೊಡಲಾಗಿದೆ.

ವಿವರಿಸಿರುವ

ನನ್ನ ಪಾಲ್ಗೊಳ್ಳುವಿಕೆಯು ಸ್ವಯಂಪ್ರೇರಿತವಾಗಿರುವುದನ್ನು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ ಮತ್ತು ನನ್ನ ವೈದ್ಯಕೀಯಆರೈಕೆಅಥವಾ ಕಾನೂನಿನ ಹಕ್ಕಿನಿಂದಯಾವುದೇ ಪರಿಣಾಮವಿಲ್ಲದೆಯೇ, ಯಾವುದೇಕಾರಣವನ್ನು ಹೇಳುವ ಮೂಲಕ ಯಾವುದೇ ಸಮಯದಲ್ಲಾದರೂ ಹಿಂಪಡೆಯಲು ನಾನು ಮುಕ್ತನಾಗಿರುತ್ತೇನೆ.

ಅಧ್ಯಯನದಿಂದ ಹಿಂತೆಗೆದುಕೊಳ್ಳುವ ಪರಿಸ್ಥಿತಿ ಉಂಟಾಗಬಹುದಾದರೆಯಾವುದೇ ಹಂತದಲ್ಲತನಿಖಾಧಿಕಾರಿಅಥವಾ ಮಾರ್ಗದರ್ಶಿಯು ನಿಮ್ಮ ಪಾಲ್ಗೊಳ್ಳುವಿಕೆಯನ್ನು ಕೊನೆಗೊಳಸಬಹುದುಎಂದು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ.

ಈ ಅಧ್ಯಯನದಿಂದ ಒದಗಿಸಿದ ಮಾಹಿತಿಗಳನ್ನು ಗೌಪ್ಯವಾಗಿಡಲಾಗುವುದು ಮತ್ತು ವೈಜ್ಞಾನಿಕ ಪ್ರಸ್ತುತಿ ಮತ್ತುಗುರುತಿನ ಮಾಹಿತಿಯಲ್ಲದೇ ಪ್ರಕಟನೆಯರೂಪದಲ್ಲ ಮಾತ್ರ ಗುಂಪು ಡೇಟಾವನ್ನು ವರದಿ ಮಾಡಲಾಗುವುದು.ಅಧ್ಯಯನದಲ್ಲ ಭಾಗವಹಿಸುವ ನನ್ನ ನಿರ್ಧಾರ ನನ್ನಚಿಕಿತ್ಸೆಯ ಮೇಲೆ ಪರಿಣಾಮ ಜೀರುವುದಿಲ್ಲ ಎಂದು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ.

ಈ ಅಧ್ಯಯನದಉಂಟಾದ ಫಲತಾಂಶದ ಬಳಕೆಯನ್ನು ನಿಬಂಧಿಸಲು ನಾನು ಸಮ್ಮತಿಸುವುದಿಲ್ಲ ಅದನ್ನು ಸೂಕ್ತ ಅಧಿಕಾರಿಗಆಗೆ ರವಾನಿಸಬಹುದು ಮತ್ತು ಪ್ರಕಟಸಬಹುದಾಗಿದೆ.

ಅಧ್ಯಯನದಲ್ಲ ಭಾಗವಹಿಸುವ ನನ್ನ ನಿರ್ಧಾರ ನನ್ನಚಿಕಿತ್ಸೆಯ ಮೇಲೆ ಪರಿಣಾಮ ಜೀರುವುದಿಲ್ಲ ಎಂದು ನಾನು ಅರ್ಥಮಾಡಿಕೊಂಡಿದ್ದೇನೆ. \_\_\_\_\_

ಸಹಿ/ಹೆಬ್ಬೆರಳು ಗುರುತಿನೊಂದಿಗೆ

ತನಿಖೆದಾರರ ಸಹಿ ಮತ್ತು ದಿನಾಂಕ

ವಿಷಯ/ಕಾನೂನು ಬದ್ದಚಿತ್ರಣದ ದಿನಾಂಕ

ಸಂಪರ್ಕ ಮಾಹಿತಿ :ತನಿಖಿದಾರರು : ಶ್ರದ್ಧಾಚಂದ್ರಶೇಖರ್

cshradha1@gmail.com

ಮಾರ್ಗದರ್ಶಕರು :ಡಾ ಕೇಶವ ಪೈ

paikeshava@gmail.com

ಆಫೀಸ್ ನಂ : 0824-2445858, - 5335

### 2. URICA – Change Assessment Scale

| University of Rhode Island | Client ID# |
|----------------------------------|--------------------------------|
| Change Assessment Scale (URICA): | Date: / /<br>Assessment Point: |
| Alcohol Version | Assessment Func |

EACH STATEMENT BELOW DESCRIBES A HOW A PERSON MIGHT FEEL WHEN STARTING THERAPY OR APPROACHING PROBLEMS IN THEIR LIVES. PLEASE INDICATE THE EXTENT TO WHICH YOU TEND TO AGREE OR DISAGREE WITH EACH STATEMENT. IN EACH CASE, MAKE YOUR CHOICE IN TERMS OF HOW YOU FEEL <u>RIGHT NOW</u>, NOT WHAT YOU HAVE FELT IN THE PAST OR WOULD LIKE TO FEEL. FOR ALL STATEMENTS THAT REFER TO YOUR "PROBLEM", ANSWER IN TERMS OF PROBLEMS RELATED TO YOUR <u>DRINKING</u>. THE WORDS "HERE" AND "THIS PLACE" REFER TO YOUR TREATMENT CENTER.

THERE ARE FIVE POSSIBLE RESPONSES TO EACH OF THE ITEMS IN THE QUESTIONNAIRE:

- 1-Strongly Disagree
- 2=Disagree
- 3-Undecided
- 4-Agree
- 5=Strongly Agree

CIRCLE THE NUMBER THAT BEST DESCRIBES HOW MUCH YOU AGREE OR DISAGREE WITH EACH STATEMENT.

| SI | ATEMENT. | Strongly<br>Disagree | Disagree | Undecided | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|---|
| 1) | I'm not the problem one. It doesn't make much<br>sense for me to consider changing. | 1 | 2 | 3 | 4 | 5 |
| 2) | I am finally doing some work on my problem. | 1 | 2 | 3 | 4 | 5 |
| 3) | I've been thinking that I might want to change something about myself. | 1 | 2 | 3 | 4 | 5 |
| 4) | At times my problem is difficult, but I'm working on it. | 1 | 2 | 3 | 4 | 5 |
| 5) | Trying to change is pretty much a waste of time<br>for me because the problem doesn't have to do<br>with me. | 1 | 2 | 3 | 4 | 5 |
| 6) | I'm hoping that I will be able to understand myself better. | 1 | 2 | 3 | 4 | 5 |
| 7) | I guess I have faults, but there's nothing that I really need to change. | 1 | 2 | 3 | 4 | 5 |
| 8) | I am really working hard to change. | 1 | 2 | 3 | 4 | 5 |
| 9) | I have a problem and I really think I should work on it. | 1 | 2 | 3 | 4 | 5 |
| 10) | I'm not following through with what I had<br>already changed as well as I had hoped, and I<br>want to prevent a relapse of the problem. | 1 | 2 | 3 | 4 | 5 |

| | | Strongly<br>Disagree | Disagree | Undecided | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|---|
| 11) | Even though I'm not always successful in<br>changing, I am at least working on my<br>problem. | 1 | 2 | 3 | 4 | 5 |
| 12) | I thought once I had resolved the problem I would be free of it, but sometimes I still find myself struggling with it. | 1 | 2 | 3 | 4 | 5 |
| 13) | I wish I had more ideas on how to solve my problem. | 1 | 2 | 3 | 4 | 5 |
| 14) | Maybe someone or something will be able to help me. | 1 | 2 | 3 | 4 | 5 |
| 15) | I may need a boost right now to help me<br>maintain the changes I've already made. | 1 | 2 | 3 | 4 | 5 |
| 16) | I may be part of the problem, but I don't really think I am. | 1 | 2 | 3 | 4 | 5 |
| 17) | I hope that someone will have some good advice for me. | 1 | 2 | 3 | 4 | 5 |
| 18) | Anyone can talk about changing; I'm actually doing something about it. | 1 | 2 | 3 | 4 | 5 |
| 19) | All this talk about psychology is boring. Why can't people just forget about their problems? | 1 | 2 | 3 | 4 | 5 |
| 20) | I'm struggling to prevent myself from having a relapse of my problem. | 1 | 2 | 3 | 4 | 5 |
| 21) | It is frustrating, but I feel I might be having a recurrence of a problem I thought I had resolved. | 1 | 2 | 3 | 4 | 5 |
| 22) | I have worries but so does the next guy. Why spend time thinking about them? | 1 | 2 | 3 | 4 | 5 |
| 23) | I am actively working on my problem. | 1 | 2 | 3 | 4 | 5 |
| 24) | After all I had done to try and change my problem, every now and then it comes back to haunt me. | 1 | 2 | 3 | 4 | 5 |

## 3. AUQ

| Date of Interview/Examination (MM/DD/YYYY): |
|---|
| Listed below are questions that ask about your feelings about drinking. The words "drinking" and "have a drink" refer to having a drink containing alcohol such as beer, wine, or liquor. Please indicate how much you agree or disagree with each of the following statements by selecting one number for each question between STRONGLY DISAGREE and STRONGLY AGREE. The closer you select a number to one end or the other indicates the strength of your disagreement or agreement. Please complete every item. We are interested in how you are thinking or feeling <u>right now</u> as you are filling out the questionnaire. |
| RIGHT NOW |
| 1. All I want to do now is have a drink. 1 [] STRONGLY DISAGREE 2 [] 3 [] 4 [] 5 [] 6 [] 7 [] STRONGLY AGREE |
| 2. I do not need to have a drink now. 1 [] STRONGLY DISAGREE 2 [] 3 [] 4 [] 5 [] 6 [] 7 [] STRONGLY AGREE |
| 3. It would be difficult to turn down a drink this minute. 1 [] STRONGLY DISAGREE 2 [] 3 [] 4 [] 5 [] 6 [] 7 [] STRONGLY AGREE |
| 4. Having a drink now would make things seem just perfect. 1 [] STRONGLY DISAGREE 2 [] 3 [] 4 [] 5 [] 6 [] 7 [] STRONGLY AGREE |
| 5. I want a drink so bad I can almost taste it. 1 [] STRONGLY DISAGREE 2 [] 3 [] 4 [] 5 [] 6 [] 7 [] STRONGLY AGREE |

| <ol><li>Nothing would be better than having a drink right now.</li></ol> | |
|---|---|
| 1 [ ] STRONGLY DISAGREE | |
| 2 []<br>3 [] | |
| 4[] | |
| 5[] | |
| 6[] | |
| 7 [ ] STRONGLY AGREE | |
| 7. If I had the chance to have a drink, I don't think I would drink 1 [] STRONGLY DISAGREE | it. |
| 2 [ ] | |
| 3[] | |
| 4[] | |
| 5[] | |
| 6 [ ]<br>7 [ ] STRONGLY AGREE | |
| /[] STRONGET AGREE | |
| 8. I crave a drink right now. | |
| 1 [ ] STRONGLY DISAGREE | |
| 2[] | |
| 3 []<br>4 [] | |
| 5[] | |
| 6[] | |
| 7 [ 1 STRONGLY AGREE | |

# 4. VAS for Coping



## 5. Directory

| | v | |
|---|---|---|
| | Patient | |
| S. No. | | Hospital No. |
| Study Code: | | Initials: |
| D.O.B: | | Gender: |
| Education: | | Occupation: |
| SES: | | Marital Status: |
| City of Residence: | | Mobile: |
| | Email: | |
| Caregiver | | |
| Name: | | Relation: |
| Education: | | Mobile: |
| | Email: | |
| (An Excel sheet will be used to record this information) | | |

## 6. Record Sheet



### 7. Randomised list of assigning conditions

11/23/2018

### A Random Permutation

from

http://www.randomization.com

Read this way ---->
9 6 8 11 12 1 19 20 14 16
18 17 3 7 13 2 15 4 5 10

To reproduce this permutation, use the seed 7244 Random permutation generated on 11/23/2018, 11:23:37 AM

### 8. Permissions

### a. URICA

### 1. University of Rhode Island Change Assessment (URICA)

Year: 1983

#### Developers:

McConnaughy, Eileen A.; Prochaska, James O.; Velicer, Wayne F.

#### Description:

The URICA is a 32-item measure that includes 4 subscales measuring the stages of change: precontemplation, contemplation, action, and maintenance. (There is also a 24-item version.) Responses are given on a 5-point Likert scale ranging from 1 (strong disagreement) to 5 (strong agreement). The subscales can be combined arithmetically (C+A+M-PC) to yield a second-order continuous Readiness to Change score that can be used to assess readiness to change at entrance to treatment.

The URICA assesses motivation for change by providing its scores on the four stages of change. Cluster analyses yielded five stages among adult outpatients entering alcoholism treatment: precontemplation, ambivalent, participation, uninvolved, and contemplation. In addition, motivation for change may be assessed using a second-order factor called Readiness to Change that seems useful at pretreatment. Clinicians may use the URICA to evaluate an individual's level of motivation for change and use this information to help guide treatment approaches. Subscale scores can be used to track shifts in attitudes related to the specific stages of change. In research, the URICA could be used to measure process and outcome variables for a variety of health and addictive behaviors. Care must be used in evaluating clients in a pre-post design since relationships among subscales shift as individuals move into action and maintenance.

The URICA can be administered in about 5-10 minutes in either a self-report or interview format.

#### **Instrument Use & Availability**

This instrument is not copyrighted. A 24item version of the URICA is also available.

#### Download the instrument:

http://adai.washington.edu/instruments/ pdf/University\_of\_Rhode\_Island\_Change \_Assessment\_258.pdf (ADAI)

#### For more information, contact:

Carlo C. DiClemente, Ph.D. Department of Psychology University of Maryland Baltimore County 1000 Hilltop Circle Baltimore, MD 21250

> Permanent URL for this page: http://bit.ly/URICA\_inst

### b. AUQ

Protocol Name from Source:

Alcohol Urge Questionnaire (AUQ)

Availability:

Publicly available

(Please Ctrl+Click on image for original source page)

MUSIC AND JPMR WITH ADS: A PILOT STUDY

| From | | Date: / / |
|---|---|---|
| Shradha Chandrasekar | | |
| Department of Psychiatry | | |
| Kasturba Medical College, | Mangalore | |
| m | | |
| To, | | |
| Re: Request for Per | mission to Inclu | ide Patient in my Study |
| Respected sir/ma'am, | | |
| Psychiatry, KMC Mangalor<br>the Use of Music and R<br>Alcohol Dependence Syn<br>alcohol dependence syndr | e, will be condu<br>elaxation Trai<br>drome: A Pilo<br>ome who have l | 09) of MSc Clinical Psychology, Department of cting a research titled 'Comparison Between ning on Craving Alcohol in Patients with t Study'. The sample consists of patients with been abstinent for at least one week of either ed, before and after, without control trial. |
| Patientcandidate to participate if | | criteria of the study and would be a good |
| The research proto and a copy of the letter fro | | proved by the Institutional Ethics Committee tached with this letter. |
| I, with this, request | your permission | n to include this patient in the research. |
| Thanking you, | | |
| Yours sincerely | | · |
| | | Guide and HOD: Dr Keshava Pai |
| Shradha Chandrasekar | | Head and Professor |
| MSc Clinical Psychology | | Dept of Psychiatry, |
| | | KMC Mangalore |
| Treating Psychiatrist: | Name: | |
| | Signature: | |
| | Date: | // |